CLINICAL TRIAL: NCT05734326
Title: Role of US Elastography Compared With FNAC in Diagnosis of Solitary Thyroid Nodule
Brief Title: Elastography and FNAC in Thyroid Nodule
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mosad Shenouda, Radiology professor Ahmed mostafa, Assiut University
Other Study IDs: Elastography & FNAC in thyroid
Record Dates: First submitted 2022-03-03; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound elastography — ultrasound elastography (USE) is emerging as a promising additional tool to discern malignant thyroid nodules, allowing increased diagnostic accuracy, Due to its ability to assess stiffness as an indicator of malignancy, USE has recently become an additional tool for thyroid nodule differentiation, in combination with conventional US and FNA [18].
  Other Names: FNAC

SUMMARY:
Evaluate the accuracy of USE in comparison with FNAC in characterization of solitary thyroid nodule and assessment the risk of malignancy

DETAILED DESCRIPTION:
Thyroid nodules occur commonly in the general population, mostly as incidental findings, with a prevalence of 19-68% at ultrasound (US) evaluation . However, although US is an established and very sensitive method for detecting thyroid nodule , it has a relatively low diagnostic performance when it comes to differentiating between benign and malignant nodules.

Therefore, when a patient presents with normal thyroid-stimulating hormone levels but US shows suspicious signs , a fine-needle aspiration biopsy (FNAB) is advised, fine-needle aspiration (FNA) is not a conclusive diagnostic method in all cases, considering its specificity, which ranges from 60 to 98%, and its variable sensitivity, which ranges from 54 to 90%, as well as the frequent eventual clinical need to repeat the test.

However, in consideration of the financial burden on health services, and to avoid unnecessary anxiety for patients, it is unrealistic to biopsy every thyroid nodule to obtain histological diagnosis.

In recent years, several studies have proposed the potential use of (US-elastography)to increase the accuracy of baseline US. Moreover, ultrasound elastography (USE) is emerging as a promising additional tool to discern malignant thyroid nodules, allowing increased diagnostic accuracy, especially in comparison with TIRADS (Thyroid Imaging Reporting and Data Systems). A firm or hard nodule consistency at palpation is associated with a high risk of malignancy. Due to its ability to assess stiffness as an indicator of malignancy, USE has recently become an additional tool for thyroid nodule differentiation, in combination with conventional US and FNA. In particular, strain ratio elastography (SRE) has shown high sensitivity and specificity, leading the EFSUMB (European Federation of Societies for Ultrasound in Medicine and Biology) to recommend that it should be part of the work-up of thyroid nodule characterization.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to radiology department presented clinically with solitary thyroid nodule .

Exclusion Criteria:

* patients previously underwent thyroid surgery
* patients with severe uncorrectable bleeding diathesis.
* Patients refused to sign consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be scanned with SWE, The thyroid gland carefully examined in the transverse and longitudinal dimensions with an 8-12 MHz linear array transducer. The shape, size, margin and echo-pattern of the lesions will be determined.then compared with FNAC results as the correct needle position inside the nodule and then in aspiration which, Finally elasticity scores and strain ratio calculations will be compared with FNAC results.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy of USE in comparison with FNAC in characterization of solitary thyroid nodule and assessment the risk of malignancy. | Base line
  Patients will be scanned with SWE The thyroid gland carefully examined in the transverse and longitudinal dimensions with an 8-12 MHz linear array transducer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gabeer, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Fresilli D, David E, Pacini P, Del Gaudio G, Dolcetti V, Lucarelli GT, Di Leo N, Bellini MI, D'Andrea V, Sorrenti S, Mascagni D, Biffoni M, Durante C, Grani G, De Vincentis G, Cantisani V. Thyroid Nodule Characterization: How to Assess the Malignancy Risk. Update of the Literature. Diagnostics (Basel). 2021 Jul 30;11(8):1374. doi: 10.3390/diagnostics11081374. PMID 34441308